CLINICAL TRIAL: NCT03244878
Title: Randomized Controlled Trial of a Culturally-adapted Version of Thrive, a Computerized Cognitive Behavior Therapy (cCBT) Program to Treat Depressive Symptoms, Syndromes, and Disorders Among Rural Montanans
Brief Title: Thrive, a Computerized Cognitive Behavior Therapy Program to Treat Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Mark B. Schure, Ph.D., Assistant Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS033017-FC
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Depressive Symptoms
Keywords: Cognitive Behavior Therapy
MeSH Terms: conditions — Depression | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either the wait-list controlled group or intervention group. Intervention period is 8 weeks. Data collection occurs at baseline, 4 weeks, and 8 weeks, with longer-term follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Thrive program (Experimental): Participants will receive access to the Thrive program for 8 weeks
  Interventions: Behavioral: Thrive
- Wait-list Control (No Intervention): Participants will have no access to the Thrive program for 8 weeks upon enrollment. They will receive a link to the NIMH website to read about information on depression.

INTERVENTIONS:
Behavioral: Thrive — A interactive computerized program using structured content of cognitive behavior therapy
  Arms: Intervention - Thrive program

SUMMARY:
This study evaluates a culturally-modified version of Thrive, a computerized Cognitive Behavior Therapy program to treat depressive symptoms, syndromes, and disorders among rural Montanans. Study participants will be randomized to either a wait-list treatment as usual or the Thrive program. After 8 weeks, the wait-list group will then receive Thrive. The primary assessment measure is the Patient Health Questionnaire-9.

DETAILED DESCRIPTION:
Montana ranks high among states on mental health disorder prevalence and low on access to mental health care. It has the highest suicide rate in the nation. Of Montana's 56 counties, 10 are classified as rural and 45 as frontier, accentuating distance challenges in accessing care. New treatment delivery modalities are needed to complement, supplement and augment traditional mental health care. With increase in access to the Internet, computer-administered Cognitive Behavior Therapy (cCBT) programs have emerged as viable approaches to effective treatment of depression.

Thrive is an interactive cCBT program with a heavy emphasis on video rather than text content that appears to improve participant engagement, a shortcoming seen in prior cCBT programs.

The goal of this project is to conduct a randomized wait-list controlled of Thrive to determine its effectiveness in reducing depressive symptom severity among Montanans, many of whom have few or no other options for mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Baseline PHQ-9 score of 5 or greater
* Montana resident
* Regular access to broadband internet (streaming capability)

Exclusion Criteria:

* No broadband internet access
* Aged 17 years or younger
* Does not have Montana residency
* Baseline PHQ-9 score of < 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | 2 weeks
  Clinical measure of depressive symptom severity. Self-reported with a score range from 0 to 3 (not at all to nearly every day)

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | 2 weeks
  Self-reported measure of anxiety symptoms with a scale from 0 to 3 (not at all to nearly every day)
Work and Social Adjustment Scale | 1 year
  Self-reported measure of a chronic condition's impact on daily work and social life with a scale of 0 to 8 (none to very severe)
Connor-Davidson Resilience Scale | 1 month
  Self-reported assessment of personal resilience with a scale of 0 to 3 (not true at all to often true)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schure M, McCrory B, Tuchscherer Franklin K, Greist J, Weissman RS. Twelve-Month Follow-Up to a Fully Automated Internet-Based Cognitive Behavior Therapy Intervention for Rural Adults With Depression Symptoms: Single-Arm Longitudinal Study. J Med Internet Res. 2020 Oct 2;22(10):e21336. doi: 10.2196/21336. PMID 33006561
- [Derived] Schure MB, Lindow JC, Greist JH, Nakonezny PA, Bailey SJ, Bryan WL, Byerly MJ. Use of a Fully Automated Internet-Based Cognitive Behavior Therapy Intervention in a Community Population of Adults With Depression Symptoms: Randomized Controlled Trial. J Med Internet Res. 2019 Nov 18;21(11):e14754. doi: 10.2196/14754. PMID 31738173

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03244878/Prot_SAP_000.pdf